CLINICAL TRIAL: NCT03470506
Title: A Study of the Relationship of Gut Microbial Composition and Stroke Outcome
Acronym: GEMSTONE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Virginia (Other)
Collaborators: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Other Study IDs: 20154
Record Dates: First submitted 2017-12-29; First posted 2018-03-20 (Actual); Last update posted 2019-11-19 (Actual); Status verified 2019-11

CONDITIONS: Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Fecal and blood samples will be collected. The biorepository will contain acute and convalescent samples: DNA (genetic and epigenetic), RNA (gene expression), serum/plasma (biomarker levels, proteomics), and fecal (microbiome) samples couple with clinical and research data.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Ischemic stroke: Diagnosed with an ischemic stroke by a Neurologist
  Interventions: Other: Stool Samples

INTERVENTIONS:
Other: Stool Samples — Stool samples will be collected at baseline and 3 months to assess differences in microbiome composition between groups

SUMMARY:
The purpose of this study is to investigate the relationship between gut microbiome (bacteria in the gut), inflammation and the injured brain. It has been established that bacteria in the gut play key roles in digestion, nutrition absorption and immune response of the entire body. Human intestinal bacteria composition in the gut has been associated with several stroke risk factors including obesity, insulin resistance, diabetes and hypertension. If we can establish a relationship between gastrointestinal microbial community composition and ischemic stroke outcomes could lead to dietary interventions in the future to improve recovery after a stroke.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women at least 18 years of age.
2. Willing and able to attend all study visits.
3. English speaking.
4. Must have had a stroke that occurred within 48 hours of admission to the Stroke Unit as determined by a neurologist.

Exclusion Criteria:

1. History of inflammatory bowel disease.
2. Receiving antibiotics within 30 days of entry into the study.
3. History of institutionalization for mental illness within the last year.
4. Unable to consent and does not have a surrogate available to consent on their behalf.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Community probability sample of adults who have suffered an ischemic stroke within 48 hours of admission to UVA
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2018-02-20 (Actual); Primary Completion 2022-01-06 (Estimated); Study Completion 2022-07-01 (Estimated)

PRIMARY OUTCOMES:
Measured differences in taxonomic make-up and the relative frequency of the gut microbial composition in relation to excellent vs. poor stroke outcome | Baseline, 3 months
  The primary outcome in this case-comparison design of those with excellent vs. non-excellent ischemic stroke outcomes at 3 months as measured by the National Institutes of Health Stroke Scale (NIHSS) is the taxonomic make up of the gut microbial composition. In other words, comprehensive microbiota survey results from 16S rRNA gene sequencing from individuals with excellent outcomes versus all other outcomes at 3 months are the outcome.

SECONDARY OUTCOMES:
Cogstate cognitive correlates and post-stroke microbial composition | Baseline, 3 months
  Descriptive analyses will be used to develop a preliminary understanding of microbiome composition in relation to measures of cognitive functioning as derived from Cogstate cognitive assessment results at baseline and 3 months post- ischemic stroke

CONTACTS AND LOCATIONS:
Overall Officials: Bradford Worrall, MD, MS, Principal Investigator — University of Virginia
Locations (2):
- United States (2):
  - University of Virginia Health System, Charlottesville, Virginia
  - Inova Health System, Fairfax, Virginia